CLINICAL TRIAL: NCT01898897
Title: Combined Anesthesia Considerations in Uro-Genital Robot Assisted Laparoscopic Surgeries: Acute Kidney Injury
Brief Title: Influence of Anesthesia Technique on Postoperative Evolution After Urogenital Surgical Interventions
Acronym: ROBOTNGAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihaly Orsolya, MD, PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Iuliu Hatieganu University
Record Dates: First submitted 2013-07-01; First posted 2013-07-15 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Anesthesia; Reaction; Adverse Effect of Other General Anesthetics; Adverse Anesthesia Outcome; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Anesthesia, Epidural; Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- robot general anesthesia (Active Comparator): General anesthesia for robot assisted laparoscopic urogenital surgery includes premedication with alprazolam (0.5 mg per os), induction with sufentanil, propofol (1-2 mg/kg), neuromuscular blocking agents (rocuronium 0.5 mg/kg) to facilitate tracheal intubation. Anesthesia is maintained with volatile agents (sevoflurane, desflurane) and reinjection of rocuronium and sufentanil as needed.
  Robotic assisted laparoscopic interventions are realised with Da Vinci surgical robot, known to assure a minimally invasive approach with good results in urologic surgery. The system consists of an ergonomic surgeon console, a patient cart with four interactive robotic arms, a 3D high resolution visualization interface and specific EndoWrist articulated tools.
  Interventions: Procedure: robot assisted laparoscopic urogenital surgery
- robot combined anesthesia (Experimental): Combined anesthesia is defined as association of epidural analgesia to general anesthesia. Epidural catheter is inserted at low thoracic level in the operation theatre before the induction of anesthesia. Correct position is verified with 15 mg bupivacaine plain 0.5%. Infusion is started after the incision at a rate of 6-8 ml/ hour.Epidural continuous infusion of local anesthetic is maintained 12 hours postoperative in the postoperative anesthesia care unit.
  Interventions: Procedure: epidural catheter insertion; Procedure: robot assisted laparoscopic urogenital surgery

INTERVENTIONS:
Procedure: epidural catheter insertion — A catheter is placed in the epidural space at thoracic level. Analgesia is realised with local anesthetics (Bupivacaine plain 0.125%), administered from the beginning of surgical intervention and 12 hours postoperative on the postoperative care unit and intensive care unit at a rate of 6-8 ml/hour.
  Other Names: peridural anesthesia and analgesia
  Arms: robot combined anesthesia
Procedure: robot assisted laparoscopic urogenital surgery — The urogenital laparoscopic surgery is assisted by DaVinci robot. The majority of interventions were prostatectomies.

SUMMARY:
The study hypothesis is that regional anesthesia offers better outcome for the patients who underwent robot assisted laparoscopic urogenital surgery.

DETAILED DESCRIPTION:
The study investigates the effect of combined anesthesia on occurrence of acute kidney injury in robot assisted laparoscopic urogenital surgery.Renal function is assessed according to the new RIFLE and AKIN criteria, and by determining serum and urinary neutrophil gelatinase associated lipocalin.

ELIGIBILITY:
Inclusion Criteria:

* signed the informed consent without previous renal function alteration respiratory and hemodynamic stability

Exclusion Criteria:

* refuse to sign the informed consent chronic or and stage renal disease severe systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 4 days
  Acute kidney injury, previously referred as acute renal failure is a serious complication of major surgery. The diagnostic of subclinical alteration of kidney function is possible with the novel biomarkers, such as neutrophil gelatinase associated lipocalin (NGAL). Modified NGAL values can be detected in patients urine and serum at 6 hours from the renal injury.
  In our study, we assessed the renal function by determining basal creatinine and follow the creatinine values 4 days postoperative. Acute kidney injury (AKI)is defined as a 0.3 mg/ml rise in serum creatinine from baseline, according to the AKIN criteria.
  NGAL is measured (with ELISA technique) at 6 hours and 12 hours from the induction of the anesthesia.
  The incidence of AKI will be compared in the different anesthesia techniques for robot assisted urogenital laparoscopic surgery.

SECONDARY OUTCOMES:
postoperative outcome | 10 days
  We study the effect of combined anesthesia (general anesthesia with epidural anesthesia and postoperative analgesia for 12 hours)on the postoperative outcome of patients who underwent robot assisted laparoscopic surgery. The endpoints that are discussed are perioperative morbidity, postoperative rehabilitation and the modification of host immune response to surgery.
  Postoperative rehabilitation is assessed by quality of recovery score (QoR-40). The modification of immune response is assessed by determining IL6, IL10 and TNFalfa levels.
  Post-prostatectomy increase in PSA (prostate specific antigen)indicates biochemic cancer recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ionescu, MD, Phd, Study Director — Iuliu Hatieganu University of Medicine
Locations (1):
- City Clinical Hospital Cluj Urology and ICU Departments, Cluj-Napoca, Cluj, Romania

REFERENCES:
- [Background] Kurosawa S, Kato M. Anesthetics, immune cells, and immune responses. J Anesth. 2008;22(3):263-77. doi: 10.1007/s00540-008-0626-2. Epub 2008 Aug 7. PMID 18685933
- [Background] Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, Collins KS; MASTER Anaethesia Trial Study Group. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet. 2002 Apr 13;359(9314):1276-82. doi: 10.1016/S0140-6736(02)08266-1. PMID 11965272
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Result] Curatolo M. Adding regional analgesia to general anaesthesia: increase of risk or improved outcome? Eur J Anaesthesiol. 2010 Jul;27(7):586-91. doi: 10.1097/EJA.0b013e32833963c8. PMID 20404731
- [Result] Wolf AR. Effects of regional analgesia on stress responses to pediatric surgery. Paediatr Anaesth. 2012 Jan;22(1):19-24. doi: 10.1111/j.1460-9592.2011.03714.x. Epub 2011 Oct 14. PMID 21999144